CLINICAL TRIAL: NCT01584726
Title: Nebulized Magnesium Sulfate in Children With Moderate to Severe Asthma Exacerbation: A Randomized, Double-Blind, Controlled Trial (RCT)
Brief Title: Nebulized Magnesium Sulfate in Children With Moderate to Severe Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #12095/12
Record Dates: First submitted 2012-04-17; First posted 2012-04-25 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
Keywords: magnesium; nebulization; asthma; sulfate; children; pediatric
MeSH Terms: conditions — Asthma | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- magnesium sulfate arm (Other): magnesium sulfate with standard therapy
  Interventions: Drug: Magnesium Sulfate
- placebo arm (No Intervention): placebo with standard therapy

INTERVENTIONS:
Drug: Magnesium Sulfate — single dose of magnesium sulfate nebulization
  Arms: magnesium sulfate arm

SUMMARY:
The purpose of this study is to investigate the use of magnesium sulfate nebulization in patient with moderate to severe asthma exacerbation in pediatric emergency.

DETAILED DESCRIPTION:
the use of magnesium sulfate nebulization in patient with moderate to severe asthma exacerbation in pediatric emergency

follow asthma severity score and length of stay

ELIGIBILITY:
Inclusion Criteria:

* Pediatric asthma patients with moderate to severe exacerbation

Exclusion Criteria:

* Known allergy to magnesium sulfate
* History of neuromuscular disease, cardiac disease, renal disease, or underlying chronic lung disease
* Use of oral steroid medication within 72 hours of presentation
* Radiographic evidence of pneumonia at presentation
* Administration of intravenous magnesium sulfate prior to study enrollment

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-03 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Would the use of nebulized magnesium sulfate in patients with moderate to severe asthma significantly reduce the time to clinical readiness for discharge? | 36 months

SECONDARY OUTCOMES:
• Would the use of nebulized magnesium sulfate in patients with moderate to severe asthma decrease admission and readmission rate, compared to placebo | 36 months
  * Would the use of nebulized magnesium sulfate in patients with moderate to severe asthma decrease PICU admission rate, compared to placebo?
  * Would the use of nebulized magnesium sulfate in patients with moderate to severe asthma improve change in asthma severity score at 4, 8, 12 hours, compared to placebo?
  * Would the use of nebulized magnesium sulfate in patients with moderate to severe asthma decrease return rate to emergency services, compared to placebo?
  * Would the use of nebulized magnesium sulfate in patients with moderate to severe asthma decrease rate of infirmray admission in follow up, compared to placebo?

CONTACTS AND LOCATIONS:
Overall Officials: KHALID AL ANSARI, MD, Principal Investigator — SENIOR CONSULTANT-HEAD OF PEDIATRIC EMERGENCY
Locations (2):
- Qatar (2):
  - Hamad Medical Corporation, Doha, Qatar
  - Pediatric Emergency Centre, Doha

REFERENCES:
- [Derived] Alansari K, Ahmed W, Davidson BL, Alamri M, Zakaria I, Alrifaai M. Nebulized magnesium for moderate and severe pediatric asthma: A randomized trial. Pediatr Pulmonol. 2015 Dec;50(12):1191-9. doi: 10.1002/ppul.23158. Epub 2015 Feb 4. PMID 25652104